CLINICAL TRIAL: NCT04366505
Title: Modification of Cue Reactivity by Neurofeedback in Human Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRR265 C04
Record Dates: First submitted 2020-03-30; First posted 2020-04-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: alcohol use disorder; mindfulness-based intervention; neurofeedback; ventral striatum
MeSH Terms: conditions — Alcoholism | interventions — Therapeutics; Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants will be allocated to one of two NFB groups (real NFB or control group) in a double-blind procedure.
  Participants of both groups will be further sub-divided into a mindfulness-based relapse prevention (MBRP) and a TAU group (single-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NFB + (MBRP) (Experimental): Neurofeedback (NFB) from target region or control region plus Mindfulness-based relapse prevention (for some)
  Interventions: Behavioral: Treatment as usual (TAU) and neurofeedback (NFB); Behavioral: mindfulness-based relapse prevention (MBRP) and NFB; Behavioral: MBT and sham NFB
- TAU and sham NFB (Active Comparator): TAU + Neurofeedback (NFB) from control region
  Interventions: Behavioral: TAU and sham NFB

INTERVENTIONS:
Behavioral: Treatment as usual (TAU) and neurofeedback (NFB) — This group will receive Treatment as usual (TAU) and neurofeedback (NFB). During NFB, participants will be asked to regulate the signal from a target brain region during the presentation of alcohol cues. The ventral striatum was chosen as target region.
  Arms: NFB + (MBRP)
Behavioral: mindfulness-based relapse prevention (MBRP) and NFB — This group will receive MBRP and neurofeedback (NFB). MBRP consists of 5 extensive sessions of a specific manualized mindfulness-based intervention for alcohol dependent patients which will be carried out by trained psychologists and psychotherapists. During NFB, participants will be asked to regulate the signal from a target brain region during the presentation of alcohol cues. The ventral striatum was chosen as a target region.
  Arms: NFB + (MBRP)
Behavioral: TAU and sham NFB — This group will receive TAU and sham NFB. Sham NFB means that the signal displayed to the participant is based on activity in a control region, the auditory cortex, which is not involved in cue reactivity.
  Arms: TAU and sham NFB
Behavioral: MBT and sham NFB — This group will receive MBRP and sham NFB. MBRP consists of 5 extensive sessions of a specific manualized mindfulness-based intervention for alcohol dependent patients which will be carried out by trained psychologists and psychotherapists. Sham NFB means that the signal displayed to the participant is based on activity in a control region, the auditory cortex, which is not involved in cue reactivity.
  Arms: NFB + (MBRP)

SUMMARY:
The project is geared towards the understanding of how to increase cognitive control over cue reactivity and drug craving.

DETAILED DESCRIPTION:
Project C04 aims at assessing the combined effect of two interventions targeting at reducing striatal cue reactivity and increasing cognitive control, namely mindfulness-based intervention and real-time fMRI neurofeedback. Firstly, the investigators will test whether a prior mindfulness-based intervention (WP1) is able to enhance the effect of rtfMRI NFB (WP2) and change the networks involved in regulation of cue reactivity by providing participants with explicit strategies. Secondly, the investigators will investigate whether this combined intervention leads to a better clinical outcome in terms of decreased heavy drinking days and a reduced sum of alcohol consumption three months later.

ELIGIBILITY:
Inclusion Criteria:

* alcohol use disorder according to DSM-5
* ability to provide fully informed consent and to use self-rating scales
* abstinent after detoxification for at least 5 days
* sufficient understanding of the German language

Exclusion Criteria:

* lifetime history of DSM-5 bipolar, psychotic disorder, or substance dependence other than alcohol or nicotine dependence
* current substance use other than nicotine and/or mild to moderate recreational use of cannabis as evidenced by positive urine test
* current threshold DSM-5 diagnosis of any of the following disorders: current (hypo)manic episode, major depressive disorder, generalized anxiety disorder, PTSD, borderline personality disorder, or obsessive compulsive disorder
* history of severe head trauma or other severe central neurological disorders (dementia, Parkinson's disease, multiple sclerosis)
* pregnancy or nursing infants
* use of medications or drugs known to interact with the CNS within the last 10 days, with testing at least four half-lives post last intake

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Neural Level: Blood Oxygen Level Dependent Signal within the ventral striatum | 3 consecutive days within up to two weeks
  Change of the ability to volitionally modulate brain activation to alcohol cues after training in the target area.
Clinical Level: Number of relapses | 3 months
  MBT and NFB will each lead to a reduced number of relapses during three months after treatment in comparison to the combination of TAU and sham NFB. The combined intervention is expected to lead to a larger reduction compared to the other groups. The investigators expect a higher number of days until relapse, a lower number of heavy drinking days and a lower amount of alcohol consumed by the participants during the follow-up period showing similar group differences.

SECONDARY OUTCOMES:
Functional changes in brain networks | up to two weeks
  Functional changes in brain networks related to cognitive control during cognitive task performance between baseline and post-neurofeedback fMRI sessions.
Drinking type | up to two weeks
  Short question on which kind of drinking type the participant identifies with the most
Form 90 (Miller, 1996) | up to two weeks
  Primary dependent measure of alcohol consumption
Baratt Impulsiveness Scale (BIS-15) (Meule et al., 2011) | up to two weeks
  Questionnaire assessing personality/behavioral construct of impulsivity. Scores range from 15 to 60. The BIS-15 has a four-point rating scale with a minimum value of 1 (1 = seldom/never) to a maximum of 4 (4 = almost always/always). Lower scores indicate less impulsivity and higher score mean more impulsivity.
Sensory Inventory (SI): self-assessment of sensory sensitivity for adults and adolescents (Zamoscik et al., 2017) | up to two weeks
  Questionnaire on self-assessment of sensory sensitivity. Minimum value: 1 representing "never". maximum value: 7 representing "almost always". Higher scores indicate higher sensitivity for sensory influences.
General depression scale (german: "Allgemeine Depressionsskala") (Radloff, 1977) | up to two weeks
  Self-assessment of depressive symptoms. minimum: 0 representing "seldom", maximum: 3 representing "mostly". Higher scores indicate stronger depression.
Positive and Negative Affect Schedule (PANAS) (Watson et al., 1988) | up to two weeks.
  measures mood/emotion. minimum: 1 representing "not at all", maximum: 5 representing "very much". Depending on the item, higher scores represent higher levels of positive affect and lower scores represent lower levels of negative affect.
Perceived Stress Scale (PSS) (Cohen et al., 1983) | up to two weeks
  measures stress. minimum: 1 representing "never". maximum: 5 representing "quite often". Higher scores indicate higher levels of perceived stress.
Behavioral Inhibition/Approach System (BIS/BAS) (Carver & White, 1994) | up to two weeks
  assessing individual differences in the sensitivity of the behavioral approach and the behavioral avoidance system.
Fagerström Test of Nicotine Dependence (Heatherton et al., 1991) | up to two weeks
  assessing nicotine dependence
Visual Craving Scale | up to two weeks
  Visual Analogue Scale for craving
Vocabulary test | Collected once during the baseline assessment
  Neuropsychological test
Dot-probe task with alcohol stimuli | Collected once during the baseline assessment
  Change in attentional bias to alcohol-related cues.
Dimensional card sorting task (Zelazo, 2006) | Collected once during the baseline assessment
  Neuropsychological test
Cue reactivity task (Vollstädt-Klein et al., 2011) | 2 timepoints: Before and after 2 weeks of neurofeedback.
  fMRI task. Change in BOLD during cue reactivity task.
Alcohol Abstinence Self-Efficacy Scale (DiClemente et al., 1994) | 2 weeks
  measure of craving. minimum: 1 representing "not at all", maximum: 5 representing "enormous". Higher scores indicate a high perceived temptation to drink.
Alcohol Urge Questionnaire (Bohn et al., 1995) | 2 weeks
  measure of craving
Alcohol Dependence Scale (Ackermann et al., 1999) | 2 weeks
  measure of craving. Range/response options vary depending on the question. Higher scores are predictive of DSM diagnosis of alcohol dependence.
German Inventory of Drinking Situations (DITS-40) (Victorio-Estrada, 1993) | 2 weeks
  measure of craving. minimum: 0 representing "never", maximum: 3 representing "almost always". Higher scores indicate a higher frequency to drink.
Craving Automated Scale for Alcohol (CASA) (Vollstädt-Klein et al., 2015) | 2 weeks
  measure of craving. minimum: 0 representing "never", maximum: 5 representing "always". Higher scores indicate automated craving.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinische Psychologie + Klinik für Abhängiges Verhalten und Suchtmedizin, Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Due to data protection rules, individual data cannot be shared. Cumulated data on the group level can be made available for meta-analyses on request.

REFERENCES:
- [Background] Anton RF, Moak DH, Latham P. The Obsessive Compulsive Drinking Scale: a self-rated instrument for the quantification of thoughts about alcohol and drinking behavior. Alcohol Clin Exp Res. 1995 Feb;19(1):92-9. doi: 10.1111/j.1530-0277.1995.tb01475.x. PMID 7771669
- [Background] DiClemente CC, Carbonari JP, Montgomery RP, Hughes SO. The Alcohol Abstinence Self-Efficacy scale. J Stud Alcohol. 1994 Mar;55(2):141-8. doi: 10.15288/jsa.1994.55.141. PMID 8189734
- [Background] Bohn MJ, Krahn DD, Staehler BA. Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcohol Clin Exp Res. 1995 Jun;19(3):600-6. doi: 10.1111/j.1530-0277.1995.tb01554.x. PMID 7573780
- [Derived] Weiss F, Aslan A, Zhang J, Gerchen MF, Kiefer F, Kirsch P. Using mind control to modify cue-reactivity in AUD: the impact of mindfulness-based relapse prevention on real-time fMRI neurofeedback to modify cue-reactivity in alcohol use disorder: a randomized controlled trial. BMC Psychiatry. 2020 Jun 16;20(1):309. doi: 10.1186/s12888-020-02717-7. PMID 32546139